CLINICAL TRIAL: NCT03002155
Title: Effects of a Community Exercise Program on Physical, Physiological, and Psychosocial Health Outcomes in People With Diabetic Foot Ulcers
Brief Title: Effects of a Exercise Program on Health Outcomes in People With Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Sara Morgan, Acting Assistant Professor, Dept. of Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 52222; P30DK017047 (NIH)
Record Dates: First submitted 2016-12-14; First posted 2016-12-23 (Estimated); Results first posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Diabetic Foot Ulcer; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus, Type 2

ARMS (2):
- Exercise (Experimental): EnhanceFitness exercise class, 1 hour, 3 times a week, duration of 12 weeks.
  Interventions: Other: EnhanceFitness community exercise program
- Control (No Intervention): Usual care.

INTERVENTIONS:
Other: EnhanceFitness community exercise program — Level I EnhanceFitness class is a seated fitness class that includes warm up, aerobics, cool down, balance training, strength training, and stretching.
  Other Names: Seated Exercise; Group exercise; Fitness program
  Arms: Exercise

SUMMARY:
People with diabetes are at risk for life altering complications, including diabetic foot ulcers. To heal a diabetic foot ulcer, people are often required to refrain from bearing weight on their affected limb for months. These long periods of non-weight bearing can result in severe physical deconditioning, putting these individuals at risk for further health decline. The goal of this pilot, randomized controlled trial is to evaluate the effects of a seated exercise program on clinically meaningful outcomes in people with diabetic foot ulcers. The long-term aim of this research is to improve overall health and quality of life in people with complications from diabetes.

DETAILED DESCRIPTION:
People with diabetes are at risk for life-altering complications and comorbidities. One of the most serious complications is a diabetic foot ulcer, which significantly increases risk for limb amputation. To heal a diabetic foot ulcer, patients are often instructed to refrain from bearing weight on the affected limb. This non-weight bearing protocol results in extended periods of inactivity that can lead to severe physical deconditioning, including diminished strength, endurance, and flexibility. EnhanceFitness, a community exercise program designed for older adults, holds classes that can be adapted for people who are non-weight bearing due to a healing foot ulcer. These exercise classes focus specifically on strength training, aerobic fitness, and stretching - activities that can counteract progressive deconditioning in people with diabetic foot ulcer. Health benefits associated with exercise in people with diabetes are well-established. However, for those experiencing declines in health and physical function because of healing protocols for a diabetic foot ulcer, the potential benefits of exercise are not yet known. The proposed project aims to address this gap in diabetes research.

The long-term goal of this research is to improve the health and quality of life of people with complications from diabetes. The specific goal of this project is to evaluate the effect of a seated community exercise program, EnhanceFitness, on clinically-meaningful outcomes in people with diabetic foot ulcers. Study investigators will recruit people with diabetic foot ulcers from local wound care clinics and randomly assign them to two groups. The first group will engage in EnhanceFitness, an existing community fitness program appropriate for people with weight-bearing restrictions due to wound-healing protocols. The second group will receive the standard of care, which does not include exercise recommendations. To assess the effectiveness of the seated exercise program, the investigators will compare important health outcomes between people with diabetic foot ulcers participating in EnhanceFitness and a control group with diabetic foot ulcers. Specifically, the investigators will assess physical and physiological outcomes, including glycated hemoglobin (HbA1c), lower-extremity strength, and wound healing. The investigators will also measure psychosocial outcomes, such as depression, perceived physical function, overall health, and self-reported ability to continue with exercise. Further, the investigators will evaluate the feasibility of conducting research assessing the effects of seated exercise in people with foot ulcers. The data collected in this pilot research will be used to apply for large, extramural funding that aims to mitigate physical deconditioning in people with diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

* 18 or more years of age
* diagnosis of type 2 diabetes
* undergoing treatment for a Wagner grade II, III, or IV diabetic foot ulcer
* able to attend regular exercise classes and two data collection sessions

Exclusion Criteria:

* medical conditions where aerobic or resistance exercise is contraindicated (e.g., uncontrolled cardiovascular problems)
* a score of less than 18 on the Montreal Cognitive Assessment indicating moderate cognitive impairment
* response from primary physician requesting that the participant not engage in exercise
* current participation in a regular exercise program (more than 30 minutes, more than 2 times a week)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-01; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara J Morgan, PhD, Principal Investigator — University of Washington
Locations (1):
- Northwest Hospital, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were assigned to study group at the time that the baseline appointment was scheduled for logistical reasons (i.e., to facilitate the identification and enrollment in a community-based exercise course if the participant was allocated to the exercise group).
  34 participants were allocated to treatment group, but only 24 attended a baseline session and consented to study participation.
Period: Overall Study
Arm/Group | Exercise | Control
Started | 10 | 14
Completed | 7 | 11
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Found to not meet inclusion criteria during baseline session data collection. | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise | Control | Total
Number analyzed (Participants) | 10 | 14 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (10.0) | 57.4 (11.8) | 58.2 (10.9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Women | 4 | 7 | 11
  Gender: Men | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 7 | 11 | 18
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 4 | 10 | 14
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 14 | 24
Time since diabetes diagnosis (self-reported) [Mean (Standard Deviation); unit: years] | 20.0 (14.8) | 19.1 (6.8) | 19.5 (11.6)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 32.7 (5.5) | 36.4 (10.8) | 34.8 (9.0)

OUTCOME MEASURES:

1. Primary Outcome: Glycated Hemoglobin (HbA1c) at 12-week Session
Description: Average blood glucose over a three-month period
Time Frame: 12 weeks post-intervention
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Exercise | Control
Number analyzed (Participants) | 7 | 11
percentage of HbA1c | 8.0 (1.7) | 7.0 (1.3)
Statistical Analysis 1: Comparison: Exercise vs Control; Test type: Superiority; p = .26, ANOVA — Not adjusted for multiple comparisons due to the pilot nature of the study, alpha level was 0.10

2. Primary Outcome: Chair Stand Test (5x Sit-to-Stand) at 12-week Session
Description: Measure of functional mobility and lower extremity strength. The 5x Sit-to-Stand test measures the total amount of time that it takes a individual to stand up and sit down in a chair five times. The individual is asked to stand up and sit down five times as quickly as they are able. The research staff started the stopwatch on "begin" and stopped timing after the individual had completed the fifth round of standing/sitting. Faster times are better, and scores are recorded in seconds.
Time Frame: 12 weeks post-intervention
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Exercise | Control
Number analyzed (Participants) | 7 | 11
seconds | 14.4 (2.8) | 17.1 (4.9)
Statistical Analysis 1: Comparison: Exercise vs Control; Test type: Superiority; p = 0.38, ANOVA

3. Secondary Outcome: PROMIS-Global at 12-week Session
Description: Patient-Reported Outcome Measurement Information System (PROMIS) Global 10-item short form. Results are reported as a T-score. PROMIS-Global is a self-reported questionnaire to assess global health. T-scores are calculated for 2 subscales- physical health and mental health. A higher T-score indicates better physical health and better mental health; a T-score of 50 indicates the general population mean with a standard deviation of 10. T-scores for physical health range from 16.2 to 67.7. T-scores for mental health range from 21.2 to 67.6.
Time Frame: 12 weeks post-intervention
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Exercise | Control
Number analyzed (Participants) | 7 | 11
T-score
  Physical Health | 47.5 (7.5) | 39.2 (6.9)
  Mental Health | 50.7 (10.0) | 45.7 (9.1)
Statistical Analysis 1: Comparison: Exercise vs Control; For PROMIS Global Physical; Test type: Superiority; p = 0.24, ANOVA
Statistical Analysis 2: Comparison: Exercise vs Control; For PROMIS Global Mental; Test type: Superiority; p = 0.80, ANOVA — p-value is interaction of group and time. Alpha level= 0.10; not adjusted for multiple comparisons (pilot study)

4. Secondary Outcome: PROMIS-Depression at 12 Weeks
Description: Patient-Reported Outcome Measurement Information System (PROMIS) Depression 4-item short form. Results are reported as a T-score. PROMIS-Depression is a self-reported questionnaire to assess depression. A higher T-score indicates greater depression; a T-score of 50 indicates the general population mean with a standard deviation of 10. T-scores range from 41.0 to 79.4 for the 4-item short form.
Time Frame: 12 weeks post-intervention
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Exercise | Control
Number analyzed (Participants) | 7 | 11
T-score | 48.4 (8.8) | 53.8 (8.7)
Statistical Analysis 1: Comparison: Exercise vs Control; Test type: Superiority; p = 0.81, ANOVA — p-value is interaction of group and time. Alpha level= 0.10; not adjusted for multiple comparisons (pilot study)

5. Secondary Outcome: PROMIS-Physical Function
Description: Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function 11-item short form. Results are reported as a T-score. PROMIS-Physical Function is a self-reported questionnaire to assess physical function. A higher T-score indicates better physical function; a T-score of 50 indicates the general population mean with a standard deviation of 10. T-scores range from 11.9 to 57.9 for the 11-item short form.
Time Frame: 12 weeks post-intervention
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Exercise | Control
Number analyzed (Participants) | 7 | 11
T-score | 44.6 (7.2) | 37.0 (3.2)
Statistical Analysis 1: Comparison: Exercise vs Control; Test type: Superiority; p = 0.03, ANOVA — p-value is interaction of group and time. Alpha level= 0.10; not adjusted for multiple comparisons (pilot study)

6. Secondary Outcome: Retention
Description: Feasibility measure- did the participant attend all study data collection sessions?
Time Frame: Through the end of study participation, approximately 12 weeks
Population: This is a feasibility measure of how many people completed the study from baseline to 12 weeks. Thus, the number of patients that completed the baseline session was used.
Measure: Count of Participants; unit: Participants
Arm/Group | Exercise | Control
Number analyzed (Participants) | 10 | 14
Participants | 7 | 11

7. Secondary Outcome: Adherence
Description: Feasibility measure- % classes attended by participants in the intervention group
Time Frame: Through the end of study participation, approximately 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of classes attended
Arm/Group | Exercise
Number analyzed (Participants) | 7
percentage of classes attended | 57.1 (28.9)

8. Secondary Outcome: EnhanceFitness Program Evaluation
Description: Feasibility measure, satisfaction with exercise program for participants in the intervention group. This satisfaction measure was designed by EnhanceFitness. It included 5 items, each item was rated by participants as 1 (not at all satisfied) to 5 (very satisfied). Responses for the five questions were summed and divided by 5. Scores ranged from 1-5, with better scored indicating higher satisfaction.
Time Frame: 12-weeks post-intervention
Population: Only participants in the exercise arm who attended at least one exercise class (n=6 out of 7 total).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise
Number analyzed (Participants) | 6
score on a scale | 4.8 (0.32)

9. Secondary Outcome: Adverse Events
Description: Feasibility measure- number of adverse events, if any, that occurred for each participant.
Time Frame: Through the end of study participation, approximately 12 weeks
Measure: Number; unit: adverse events
Arm/Group | Exercise | Control
Number analyzed (Participants) | 7 | 11
adverse events | 0 | 0

10. Other Pre Specified Outcome: Recruitment
Description: Feasibility measure- were overall recruitment targets reached? This feasibility measure will be assessed for the overall study and not for each participant.
Time Frame: At the completion of the 2-year study
Population: 34 is the number randomized to group; 40 is the number that we targeted for this study
Measure: Count of Participants; unit: Participants
Groups:
- Overall Sample: All of the participants who were randomized to group out of the total number targeted for this study
Arm/Group | Overall Sample
Number analyzed (Participants) | 40
Participants | 34

ADVERSE EVENTS:
Time Frame: 12 weeks (the duration of a participant's time in the study.
Arm/Group | Exercise | Control
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/11
Other Adverse Events (participants affected / at risk) | 0/7 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/55/NCT03002155/Prot_SAP_000.pdf